CLINICAL TRIAL: NCT04042038
Title: Neural Predictors and Neural Changes Associated With Cognitive Behavior Therapy for Obssesive Compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); FIDMAG Germanes Hospitalàries (Other)
Responsible Party: Principal Investigator, Carles Soriano Mas, Principal Investigator, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HCB/2018/0681
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
Keywords: Obsessive compulsive disorder; Intensive cognitive-behavioral therapy; Neuroimaging; Response prediction; Response mechanisms; Functional magnetic resonance imaging
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Two separate (but methodologically identical) RCTs will be conducted, one in a sample of children/adolescents with OCD (study 1) and another in a sample of adults with OCD (study 2). Within each study, one group of age and gender-matched healthy controls will also serve as a comparison group at baseline (clinical and neuroimaging assessment). Within each study, after baseline assessment, OCD participants will be randomized to either intensive CBT or waiting list for one month. Then, OCD participants will be assessed again (clinical and neuroimaging assessment).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT (Experimental): Intensive CBT (20 sessions in 1 month)
  Interventions: Behavioral: Cognitive-behavior therapy (psychological treatment)
- Waiting-list (No Intervention): Waiting-list

INTERVENTIONS:
Behavioral: Cognitive-behavior therapy (psychological treatment) — Participants will receive up to 20 hours of manualized and structured CBT based on exposure and response prevention by experienced clinicians
  Arms: CBT

SUMMARY:
The goals of the project are 1) to understand what are the neural mechanisms involved in the psychological treatment of obsessive-compulsive disorder (OCD) in children/adolescents and adults, 2) to assess potential differences in the neural mechanisms involved in the psychological treatment of OCD between children/adolescents and adults, and 3) to assess the effectiveness of intensive CBT for children/adolescents and adults with OCD.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a frequent and disabling disorder. Cognitive-behavior therapy (CBT) is the best treatment option available for OCD, although it achieves optimum results in less than half of the patients. The investigators will investigate the main neural circuits that predict CBT outcome in OCD and the neural changes associated with CBT in two separate randomized controlled trials (RCTs), one in an adult sample and another in a pediatric sample. In this two RCTs, OCD participants will be randomized to either intensive CBT (20 sessions in 1 month) by a experienced clinician or a waiting-list control (WLC) and will be assessed (by a blind assessor) and scanned before and after CBT. Patients will be offered CBT if they have been randomized to the WLC. At baseline, the investigators will also compare OCD patients with a group of healthy controls (HC). Secondary goals of the project include 1) assessing potential differences between children/adolescents and adults in the neural mechanisms involved in CBT for OCD; 2) assess the effectiveness of intensive CBT for children/adolescents and adults.

ELIGIBILITY:
Inclusion Criteria: (same for Study 1 and Study 2):

1. Principal diagnosis of OCD;
2. Y-BOCS or CYBOCS ≥ 16).
3. No current psychotropic medication (except benzodiacepines for sleep). 4 ) Age between 8 and 17 years (Study 1) and between 18 and 60 years (Study 2).

Exclusion Criteria: (same for Study 1 and Study 2

1. Current major depression or current/past psychosis, bipolar disorder or substance abuse.
2. Developmental disorders (including autistic spectrum disorders).
3. To be pregnant or during breastfeeding
4. Current CBT; nt.
5. Any severe medical disorder ;
6. Any contraindication for neuroimaging

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale | Change from baseline to post-treatment (1 month)
  The Yale-Brown Obsessive-Compulsive Scale evaluates the severity of Obsessive Compulsive Disorder symptoms in adults. The scale is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms) (total range, 0 to 40), with separate subtotals for severity of obsessions and compulsions.
Children´s Yale-Brown Obsessive-Compulsive Scale | Change from baseline to post-treatment (1 month)
  The Children´s Yale-Brown Obsessive-Compulsive Scale evaluates the severity of Obsessive Compulsive Disorder symptoms in children/adolescents. The severity of the obsessions is rated on five Severity Items for Obsessions. Each of these five items is rated on a 5-point, ordinal scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = extreme. These values are anchored by a description for each score. The Obsessions Severity Score is obtained by adding the scores for items 1 through 5 (range = 0 to 20).
  There are five comparable Severity Items for Compulsions (items 6 through 10), which are also scored from 0 to 4. The Compulsions Severity Score is obtained by adding the scores of items 6 through 10 (range = 0 to 20). Summing the scores for all 10 items yields the CY-BOCS Total score (range = 0 to 40).

SECONDARY OUTCOMES:
Obsessive-Compulsive Inventory-Revised | Change from baseline to post-treatment (1 month)
  Obsessive-Compulsive Inventory-Revised is a self-report scale for assessing symptoms of Obsessive-Compulsive Disorder in adults. It consists of 18 questions that a person endorses on a 5-point Likert scale. Scores are generated by adding the item scores. The possible range of scores is 0-72. Mean score for persons with OCD is 28.0 (SD = 13.53). Recommended cutoff score is 21, with scores at or above this level indicating the likely presence of OCD.
Obsessive Compulsive Inventory-Child Version | Change from baseline to post-treatment (1 month)
  Questionnaire assessing severity of obsessive-compulsive disorder symptoms children/adolescents. It is a 21-item self-report questionnaire, based on the 42-item adult version. Items are scored on a 3-point Likert scale. The measure is designed to evaluate obsessive-compulsive disorder in children between 7 and 17 years old. The total ranges from 0 to 42 points.
Children's Depression Inventory | Change from baseline to 1 month.
  The Children's Depression Inventory is a psychological assessment that rates the severity of symptoms related to depression or dysthymic disorder in children and adolescents. It is a 27-item scale that is self-rated and symptom-oriented. The 27 items on the assessment are grouped into five major factor areas. Patients rate themselves based on how they feel and think, with each statement being identified with a rating from 0 to 2.
Spence Children's Anxiety Scale | Change from baseline to 1 month
  The Spence Children's Anxiety Scale is a psychological questionnaire designed to identify symptoms of various anxiety disorders, specifically social phobia, obsessive-compulsive disorder, panic disorder/agorophobia, and other forms of anxiety, in children and adolescents between ages 8 and 15. There are 45 questions evaluating the frequency of certain anxiety symptoms, measured on a 0-3 scale from "never," "sometimes," often," to "always." A maximum score of 114 is possible on the child and parent-reported, and there are six subscales calculated within the final score. The total score is interpreted in different ways depending on the child's age and gender. For boys and girls ages 8-11, a total score of 40 and above or 50 and above is classified as elevated levels of anxiety, respectively. For boys and girls ages 12-15, a total score of 33 and above or 39 and above is classified as elevated, respectively.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - IDIBELL, L'Hospitalet de Llobregat, Barcelona
  - FIDMAG Germanes Hospitalàries, Sant Boi de Llobregat, Barcelona
  - IDIBAPS, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hermida-Barros L, Garcia-Delgar B, Lera-Miguel S, Forcadell E, Moreno E, Prime-Tous M, Jaurrieta N, Segu X, Vilajosana E, Soriano-Mas C, de la Cruz LF, Vieta E, Radua J, Lazaro L, Fullana MA. Concentrated Cognitive-Behavior Therapy for Unmedicated Children and Adolescents With Obsessive-Compulsive Disorder in Routine Clinical Care: A Randomized Controlled Trial With a 6-Month Naturalistic Follow-up. Behav Ther. 2025 Jul;56(4):799-811. doi: 10.1016/j.beth.2025.01.001. Epub 2025 Jan 13. PMID 40541379